CLINICAL TRIAL: NCT02301429
Title: Model 20105 Lead Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low implant success rate(46%). For the successfull implants, 3month FU and available electrical data showed an increase in threshold values for the left atrium
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LV DDD
Record Dates: First submitted 2014-10-20; First posted 2014-11-25 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Sick Sinus Node Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Model 20105 (Experimental): Receiving the model 20105 Lead
  Interventions: Device: Model 20105

INTERVENTIONS:
Device: Model 20105 — implant and follow-up of study device

SUMMARY:
The purpose of this study is to evaluate the implant procedure and feasibility of a new lead developed to pace and sense the left chambers of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Cardiac pacing indication for sinus node dysfunction (dual chamber pacemaker)
* Subject has signed and dated the study-specific informed consent form
* Subject is 18 years of age or older
* Subject is willing, able and committed to participate in Baseline and Follow-up and study procedures for the full length of the study

Exclusion Criteria:

* Subject is indicated for BiV pacemaker or ICD
* Subject is pacing dependent
* Subject has a previous Pacemaker System
* Subject has known coronary venous vasculature that is inadequate for lead placement
* Subject has unstable angina pectoris or has had an acute myocardial infarction (MI) within the last month
* Subject has had a coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past three months
* Subject is not in sinus rhythm at implant
* Subject has had a heart transplant (patients waiting for heart transplants are allowed in the study)
* Subject has known renal insufficiency that would prevent them from receiving an occlusive venogram during the implant procedure
* Subject is contraindicated for <1mg dexamethasone acetate
* Subject is enrolled in any concurrent drug and/or device study that may confound the results of this study
* Subject has a terminal illness and is not expected to survive more than 6 months
* Subject is a pregnant woman or woman of childbearing potential not on adequate birth control.
* Subject is employed by Medtronic or by the department of any of the investigators or is a close relative of any of the investigators.
* Legal incapacity or evidence that a subject cannot understand the purpose and risks of the study
* Subject meets exclusion criteria required by local law.
* Subject is unable to tolerate an urgent thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- London Teaching Hospital, London, Canada
- Reinier de Graaf Hospital, Delft, Netherlands
- NUHCS, National University Hospital, Singapore, Singapore
- Milpark hospital, Johannesburg, South Africa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Model 20105
Started | 16
Completed | 13
Not Completed | 3
Not completed — not acceptable vascular anatomy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Model 20105
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
QRS duration [Mean (Standard Deviation); unit: msec] | 108.7 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: All Implant Procedure and Lead Related Adverse Events Will be Collected During the First Month Post Implant and Analyzed.
Description: All Implant procedure and lead related adverse events will be collected during the first month post implant and analyzed.
Time Frame: 1 month
Population: all subject who underwent a Model 20105 Lead implant attempt are considered in this analysis
Measure: Number; unit: Adverse Events
Arm/Group | Model 20105
Number analyzed (Participants) | 13
Adverse Events | 3

ADVERSE EVENTS:
Arm/Group | Model 20105
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 20105 (N=13)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 1 (1)
Iatrogenic pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Coronary Artery Stent Insertion (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 20105 (N=13)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 1 (1)
Atrioventricular nodal reentrant tachycardia (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days